CLINICAL TRIAL: NCT06180447
Title: Peri-conceptional or Pregnancy Exposure of Vaccination and the Risk of Adverse Pregnancy Outcomes
Status: Active, not recruiting | Type: Observational
Sponsor: Sun Xin (Other)
Responsible Party: Sponsor-Investigator, Sun Xin, professor; director, West China Hospital
Organization: West China Hospital (Other)
Other Study IDs: Vaccine registry study
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Vaccine Adverse Reaction
Keywords: Vaccine; birth defect; adverse pregnancy outcomes
MeSH Terms: conditions — Congenital Abnormalities | interventions — Hepatitis B Vaccines; Rabies Vaccines; Papillomavirus Vaccines; Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Biological: Hepatitis B vaccine, rabies vaccine, HPV vaccine, influenza vaccine — Exposure was defined as use of the vaccine 90 days before the last menstrual period and during pregnancy.

SUMMARY:
Uing data from a population based cohort in China, we will conduct retrospective cohort study to evaluate the risk of vaccine (e.g., HPV/influenza/rabies vaccine) administered during pregnancy (especially during first trimester) for adverse pregnancy outcomes (e.g., birth defects, preterm birth and low birth weight)

DETAILED DESCRIPTION:
We will develop a vaccination cohort by linking population-based pregnancy registries (i.e., REPRESENT) with population-based vaccine databases.

The researchers will use data from this cohort to examine vaccine use 90 days before the last menstrual period and throughout pregnancy. This study will investigate whether maternal vaccination during pregnancy is associated with the risk of adverse pregnancy outcomes. Poisson regression based on propensity scores will be used to estimate the relative risk. To ensure the robustness of the results, the researchers will perform several sensitivity analyses and negative control analyses, such as the risk of adverse pregnancy outcomes in pregnant women who have been vaccinated several times and pregnant women who have been vaccinated in mid and late pregnancy as negative control groups.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women in Xiamen who registry in our database.

Exclusion Criteria:

* Pregnant women who were lost to follow-up. Pregnant women exposed to related factors of known congenital malformation.

Ages: 14 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For women who are pregnant during the study period, the exposed population is pregnant women who have been vaccinated during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 150000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Birth defects | From pregnancy to 42 days after delivery
  BDs were defined as any prenatal malformation (including structural, functional, or metabolic disorders) diagnosed through systematic ultrasound or genetic testing during pregnancy and any malformation diagnosed by clinicians within 42 days of birth，which were coded according to the International Classification of Diseases, Tenth Revision (ICD-10) (Q00-Q99).

SECONDARY OUTCOMES:
Incidence of Adverse pregnancy outcomes | From pregnancy to 42 days after delivery
  Including gestational diabetes, fetal distress, premature rupture of membranes, low birth weight and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Sun, PhD, Study Chair — Chinese Evidence-based Medicine Center, West China Hospital of Sichuan University
Locations (1):
- The West China Hospital of Sichuan university, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
The datasets are not publicly available, but are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Guo J, Zhao P, Liu C, Liao M, Chen J, Ren Y, Yao G, Qian Y, Rong B, Qi H, Chen M, Zou K, Xiong Y, Sun X, Tan J. Peri-Conception Human Papillomavirus Vaccination Exposure and Risk of Birth Defects: A Population-Based Retrospective Cohort Study. Pharmacoepidemiol Drug Saf. 2025 Oct;34(10):e70222. doi: 10.1002/pds.70222. PMID 40984047